CLINICAL TRIAL: NCT01939678
Title: Characterization and Role of Mutations in Sodium-phosphate Cotransporters in Patients With Calcific Aortic Valve Disease
Status: Terminated | Type: Observational
Why Stopped: Enrollment lower than expected
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Ole Frobert, MD, PhD, MD, PhD, Region Örebro County
Other Study IDs: 2012-12
Record Dates: First submitted 2013-08-27; First posted 2013-09-11 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloodsamples and Aortic valve samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate whether mutations in genes coding for Na/Pi-cotransporters are associated with aortic valve calcification. A patient population with premature aortic valve calcification treated with aortic valve replacement will be screened for mutations in these specific genes. Furthermore, aortic valve tissue received from the operations, will be examined for the presence of Na/Pi-cotransporters, and for molecular characterization of the transporters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aortic valve calcification that will be treated with an aortic valve replacement.
* Age ≤ 65 years.
* Signed and dated informed consent.

Exclusion Criteria:

* Inability to provide informed consent
* Earlier radiation therapy of the thorax
* Severe renal disease (patients in treatment with dialysis)

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with aortic valve calcification that will be treated with an aortic valve replacement
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-09; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Mutations in sodium-phosphate cotransporters in patients with calcific aortic valve disease | At the time of aortic valve replacement
  Mutations in genes coding for Na/Pi-cotransporters

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Orebro University Hospital, Örebro, Sweden